CLINICAL TRIAL: NCT05007041
Title: Safety of Simultaneous Vaccination With Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Inactivated Influenza Vaccine (aIIV4)
Brief Title: Simultaneous RZV and aIIV4 Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00108456
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Pain; Quality of Life; Injection Site Reaction; Adverse Drug Event
Keywords: influenza vaccine; fever following vaccination; pain following vaccination; quality of life; Zoster Vaccine Recombinant, Adjuvanted (RSV) (SHINGRIX®); Quadrivalent Influenza Vaccine, Adjuvanted (FLUAD®); Fluzone(®) High-Dose Quadrivalent
MeSH Terms: conditions — Pain; Injection Site Reaction; Drug-Related Side Effects and Adverse Reactions; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, study coordinators, and investigators will be blinded to the type of influenza vaccine administered in conjunction with the Recombinant Zoster Vaccine, Adjuvanted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine (FLUAD®) (Active Comparator): In this study arm, subjects will receive Dose 1 of RZV (SHINGRIX®) and Dose 1 of the adjuvanted influenza vaccine (FLUAD® Quadrivalent) simultaneously during Visit 1 and Dose 2 of RZV (SHINGRIX®) during Visit 6.
  Interventions: Biological: FLUAD® Quadrivalent; Biological: SHINGRIX®
- Zoster Vaccine Recombinant (RZV) and High-Dose Quadrivalent Influenza Vaccine (Fluzone®) (Active Comparator): In this study arm, subjects will receive Dose 1 of RZV (SHINGRIX®) and Dose 1 of the (Fluzone® HD Quadrivalent) influenza vaccine simultaneously during Visit 1 and Dose 2 of RZV (SHINGRIX®) during Visit 6.
  Interventions: Biological: Fluzone® High-Dose Quadrivalent; Biological: SHINGRIX®

INTERVENTIONS:
Biological: FLUAD® Quadrivalent — Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  Other Names: Influenza Vaccine, Adjuvanted (Quadrivalent); aIIV4
  Arms: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine (FLUAD®)
Biological: Fluzone® High-Dose Quadrivalent — Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  Other Names: High-Dose Quadrivalent Influenza Vaccine; HD-IIV4
  Arms: Zoster Vaccine Recombinant (RZV) and High-Dose Quadrivalent Influenza Vaccine (Fluzone®)
Biological: SHINGRIX® — Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  Other Names: Zoster Vaccine Recombinant, Adjuvanted (RZV)

SUMMARY:
The overall aim of the study is to compare the safety of simultaneous Zoster Vaccine Recombinant, Adjuvanted (RZV) (SHINGRIX®) and Quadrivalent Influenza Vaccine, Adjuvanted (FLUAD®) versus simultaneous Zoster Vaccine Recombinant, Adjuvanted (RZV) (SHINGRIX®) and Fluzone® High-Dose Quadrivalent vaccine in persons age ≥65 years. A prospective, randomized, blinded clinical trial that will be conducted during the 2021/2022 and 2022/2023 influenza seasons. Over the course of these two influenza seasons, approximately 220 older adults will be enrolled at Duke University Medical Center, and 180 older adults at Johns Hopkins University Medical Center. Eligible subjects will be randomized to receive either simultaneous RZV/FLUAD® or RZV/Fluzone® High-Dose vaccines. All subjects will be assessed for 7 days post-injection and safety and tolerability compared between the two groups. Serious adverse events and adverse events of clinical interest will be assessed 42 days post-vaccination and compared between the two groups. Health-related quality of life will be assessed pre-vaccination Day 1 through Day 8. Serious Adverse Events and Adverse Events of Clinical Interest were also assessed throughout the study period.

DETAILED DESCRIPTION:
Intention-to-Treat (ITT) Population: Defined as all subjects who are randomized and vaccinated.

Modified Intention-to-Treat (mITT) Population: Defined as all subjects who are randomized, vaccinated, and provide at least one day of complete data on the symptom diary.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 65 years
2. Intention of receiving IIV and RZV based on ACIP-CDC guidelines
3. Able to speak English
4. Willing to provide written informed consent
5. Living in the community
6. Intention of being available for entire study period and complete all relevant study procedures, including follow-up phone calls and clinic visits.
7. If HIV positive, HIV should be clinically stable.

Exclusion Criteria:

1. IIV or recombinant influenza vaccine (RIV) receipt during the respective 2021-2022 or 2022-2023 influenza season prior to study enrollment
2. Prior receipt of recombinant zoster vaccine (SHINGRIX®)
3. For non-COVID-19 Vaccines:

   * Receipt of any inactivated vaccine within 2 weeks prior to enrollment in this study
   * Receipt of any live vaccine within 4 weeks prior to enrollment in this study
   * Planning receipt of any non-COVID-19 vaccine during the entire period
4. For COVID-19 Vaccines:

   * Receipt of COVID-19 vaccine within 2 weeks prior to enrollment in this study. For those who have initiated a COVID-19 vaccine series, enrollment is not allowed until 2 weeks after the final dose of a COVID-19 vaccine is completed.
   * Planning receipt of a COVID-19 vaccine within 2 weeks after administration of study influenza and first dose recombinant zoster study vaccines.
5. Have acute illness or exacerbation of chronic illness within 72 hours of study vaccination
6. Hospitalization within the last 30 days for any reason
7. History of febrile illness (> 100.0°F or 37.8°C) within the past 24 hours prior to IIV administration
8. Has immunosuppression as a result of an underlying illness or treatment, or use of chemotherapy or radiation therapy within the preceding 12 months
9. Has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) *Participants with a history of malignancy may be included if, after previous treatment by surgical excision, chemotherapy or radiation therapy, the participant has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure
10. A history of autoimmune disease, that requires immunosuppressive agents or any other chronic medical condition considered clinically significant by the investigator
11. Use of chronic oral or intravenous administration (≥14 days) of immunosuppressive doses of steroids, i.e., prednisone >10 mg per day, immunosuppressants or other immune-modifying drugs within 30 days of starting this study. (Use of topical, nasal, or inhaled steroids is permitted)
12. Thrombocytopenia, bleeding disorder, or anticoagulant use contraindicating intramuscular injection (a daily aspirin may be acceptable)
13. Contraindication to IIV receipt including history of severe allergic reaction after a previous dose of any influenza vaccine; or to a vaccine component, including egg protein
14. Contraindication to RZV including history of a severe allergic reaction to any component of the RZV vaccine (including saponin or polysorbate 80) or to dose 2 of RZV
15. History of Guillain-Barré syndrome
16. History of Hepatitis C or active Hepatitis B
17. Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
18. Dementia, any cognitive condition, or substance abuse that could interfere with study compliance
19. Anyone who is already enrolled or plans to enroll in another clinical trial with an investigational product within 28 days of vaccine receipt. Co-enrollment in observational or behavioral intervention studies are allowed at any time while enrollment in a clinical trial involving an investigational product (other than vaccine) may occur after 28 days following vaccine receipt
20. Any condition which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives
21. Anyone who is a relative of any research study personnel
22. Anyone who is an employee of any research study personnel

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 267 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Schmader, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmader KE, Walter EB, Talaat KR, Rountree W, Poniewierski M, Randolph E, Leng SX, Wunderlich B, McNeil MM, Museru O, Broder KR. Safety of Simultaneous Vaccination With Adjuvanted Zoster Vaccine and Adjuvanted Influenza Vaccine: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2440817. doi: 10.1001/jamanetworkopen.2024.40817. PMID 39446325
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine: In this study arm, subjects will receive Dose 1 of RZV (SHINGRIX®) and Dose 1 of the quadrivalent adjuvanted influenza vaccine (FLUAD® Quadrivalent) simultaneously during Visit 1 and Dose 2 of RZV (SHINGRIX®) during Visit 6.
  FLUAD® Quadrivalent: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  SHINGRIX®: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
- Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine: In this study arm, subjects will receive Dose 1 of RZV (SHINGRIX®) and Dose 1 of the (Fluzone® HD Quadrivalent) influenza vaccine simultaneously during Visit 1 and Dose 2 of RZV (SHINGRIX®) during Visit 6.
  Fluzone® HD Quadrivalent: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  SHINGRIX®: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
Period: Overall Study
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Started | 130 | 137
Completed | 130 | 136
Not Completed | 0 | 1
Not completed — Missing Diary Entries | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine | Total
Number analyzed (Participants) | 130 | 137 | 267
Age, Customized [Count of Participants; unit: Participants]
  65-69 years | 44 | 48 | 92
  70 or more years | 86 | 89 | 175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 69 | 130
  Male | 69 | 68 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 128 | 134 | 262
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Only | 123 | 124 | 247
  Black Only | 7 | 12 | 19
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Local or Systemic Reactogenicity Event After Dose 1 of RZV (SHINGRIX®) in Each Study Group
Description: Modified Intention-to-Treat (mITT) Population
Time Frame: Up to 8 days post-vaccination
Population: Modified Intention-to-Treat (mITT) Population: All subjects who are randomized, vaccinated (received at least one study vaccine), and provided at least one day of complete data on the symptom diary.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 130 | 136
Participants
  No | 115 | 119
  Yes | 15 | 17
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; The null hypothesis is simultaneous vaccination with RZV and allV4 is inferior (i.e., RZV and allV4 will have a higher proportion) to RZV and HD-IIV4 with regard to the proportion of adults with at least one severe (Grade 3) solicited local or systemic reactogenicity event on days 1-8 after RZV dose; Test type: Non-Inferiority — The one-sided non-inferiority test with the alpha level set at 0.025 and non-inferiority margin of 10%, stratified by site; p = 0.0037, Difference in proportions; The upper bound of a site-stratified Newcombe binomial confidence interval with Cochran-Mantel-Haenszel weighting of the difference was used; Difference in proportions = -0.96, 95% CI 2-sided [-8.94 to 7.10]

2. Primary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Local or Systemic Reactogenicity Event After Dose 1 of RZV (SHINGRIX®) in Each Study Group - Ages 65-69
Description: Modified Intention-to-Treat (mITT) Population
Time Frame: Up to 8 days post-vaccination
Population: Modified Intention-to-Treat (mITT) Population: All subjects ages 65-69 who are randomized, vaccinated (received at least one study vaccine), and provided at least one day of complete data on the symptom diary.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 44 | 48
Participants
  No | 41 | 41
  Yes | 3 | 7
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Other — Difference in proportions; Difference in proportions = -7.77, 95% CI 2-sided [-20.22 to 4.69]

3. Primary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Local or Systemic Reactogenicity Event After Dose 1 of RZV (SHINGRIX®) in Each Study Group - Ages 70 and Older
Description: Modified Intention-to-Treat (mITT) Population
Time Frame: Up to 8 days post-vaccination
Population: Modified Intention-to-Treat (mITT) Population: All subjects ages 70 or older who are randomized, vaccinated (received at least one study vaccine), and provided at least one day of complete data on the symptom diary.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 86 | 88
Participants
  No | 74 | 78
  Yes | 12 | 10
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Other — Difference in proportions; Difference in proportions = 2.59, 95% CI 2-sided [-7.29 to 12.47]

4. Secondary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Local Reactogenicity Event After Dose 1 of RZV (SHINGRIX®) in Each Study Group
Description: Modified Intention-to-Treat (mITT) Population
Time Frame: Up to 8 days post-vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 130 | 136
Participants
  No | 122 | 130
  Yes | 8 | 6
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Number of Participants With at Least One Severe (Grade 3) Solicited Local Reactogenicity Event After SHINGRIX® Dose 1 in Each Study Group; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0031, Difference in proportions — The upper bound of a site-stratified Newcombe binomial confidence interval with Cochran-Mantel-Haenszel weighting of the difference was used; Difference in proportions = 1.74, 95% CI 2-sided [-4.04 to 7.77]

5. Secondary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Local Reactogenicity Event After Dose 1 of RZV (SHINGRIX®)in Each Study Group - Ages 65-69
Description: Modified Intention-to-Treat (mITT) Population
Time Frame: Up to 8 days post-vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 44 | 48
Participants
  No | 44 | 45
  Yes | 0 | 3
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Other — Difference in proportions; Difference in proportions; Difference in proportions = -6.25, 95% CI 2-sided [-13.10 to 0.60]

6. Secondary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Local Reactogenicity Event After Dose 1 of RZV (SHINGRIX®) in Each Study Group - Ages 70 and Older
Description: Modified Intention-to-Treat (mITT) Population
Time Frame: Up to 8 days post-vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 86 | 88
Participants
  No | 78 | 85
  Yes | 8 | 3
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Other — Difference in proportions; Difference in proportions; Difference in proportions = 5.89, 95% CI 2-sided [-1.32 to 13.11]

7. Secondary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Systemic Reactogenicity After Dose 1 of RZV (SHINGRIX®) in Each Study Group
Description: Modified Intention-to-Treat (ITT) Population. Two subjects in the High-dose Quadrivalent Influenza arm reported local and systemic grade 3 events
Time Frame: Up to 8 days post-vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 130 | 136
Participants
  No | 123 | 123
  Yes | 7 | 13
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Difference in proportions; [statistical method as in outcome 1, analysis 1]; Difference in proportions = -4.17, 95% CI 2-sided [-10.90 to 2.47]

8. Secondary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Systemic Reactogenicity After Dose 1 of RZV (SHINGRIX®) in Each Study Group - Ages 65-69
Description: as for outcome 7
Time Frame: Up to 8 days post-vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 44 | 48
Participants
  No | 41 | 42
  Yes | 3 | 6
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Other — Difference in proportions; Difference in proportions; Difference in proportions = -5.68, 95% CI 2-sided [-17.64 to 6.28]

9. Secondary Outcome: Number of Participants With at Least One Severe (Grade 3) Solicited Systemic Reactogenicity After Dose 1 of RZV (SHINGRIX®) in Each Study Group - Ages 70 and Older
Description: Modified Intention-to-Treat (ITT) Population
Time Frame: Up to 8 days post-vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 86 | 88
Participants
  No | 82 | 81
  Yes | 4 | 7
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Other — Difference in proportions; Difference in proportions; Difference in proportions = -3.30, 95% CI 2-sided [-10.50 to 3.89]

10. Secondary Outcome: Number of Participants With at Least One Adverse Event of Clinical Interest After Dose 1 of RZV (SHINGRIX®) in Each Study Group
Description: Intention-to-Treat (ITT) Population
Time Frame: Up 43 days post-vaccination
Population: ITT Population: All subjects who are randomized and vaccinated (received at least one study vaccine).
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 130 | 137
Participants
  No | 130 | 136
  Yes | 0 | 1
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Other — Difference in proportions; Difference in proportions; Difference in proportions = -0.73, 95% CI 2-sided [-2.16 to 0.70]

11. Secondary Outcome: Number of Participants With at Least One Serious Adverse Event After Dose 1 of RZV (SHINGRIX®) in Each Study Group
Description: Intention-to-Treat (ITT) Population
Time Frame: Up 43 days post-vaccination
Population: ITT Population: All subjects who are randomized and vaccinated (received at least one study vaccine).
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 130 | 137
Participants
  No | 129 | 132
  Yes | 1 | 5
Statistical Analysis 1: Comparison: Zoster Vaccine Recombinant (RZV) and Quadrivalent Adjuvanted Influenza Vaccine vs Zoster Vaccine Recombinant (RZV) and High-dose Quadrivalent Influenza Vaccine; Test type: Other — The proportion and 95% exact binomial confidence interval between vaccine groups; Difference in proportions; Difference in proportions = -2.88, 95% CI 2-sided [-6.36 to 0.60]

ADVERSE EVENTS:
Time Frame: Participants were followed through Day 43 after each dose of SHINGRIX for adverse events and adverse events of clinical interest. Participants were followed through the entire study period (up to 110 days) for serious adverse events.
Groups:
- Recombinant Zoster Vaccine (RZV) and Quadrivalent Adjuvanted Influenza Vaccine: In this study arm, subjects will receive Dose 1 of RZV (SHINGRIX®) and Dose 1 of the quadrivalent adjuvanted influenza vaccine (FLUAD® Quadrivalent) simultaneously during Visit 1 and Dose 2 of RZV (SHINGRIX®) during Visit 6.
  FLUAD® Quadrivalent: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  SHINGRIX®: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
- Recombinant Zoster Vaccine (RZV) and High-Dose Quadrivalent Influenza Vaccine: In this study arm, subjects will receive Dose 1 of RZV (SHINGRIX®) and Dose 1 of the (Fluzone® HD Quadrivalent) influenza vaccine simultaneously during Visit 1 and Dose 2 of RZV (SHINGRIX®) during Visit 6.
  Fluzone® HD Quadrivalent: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  SHINGRIX®: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
Arm/Group | Recombinant Zoster Vaccine (RZV) and Quadrivalent Adjuvanted Influenza Vaccine | Recombinant Zoster Vaccine (RZV) and High-Dose Quadrivalent Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/137
Serious Adverse Events (participants affected / at risk) | 4/130 | 5/137
Other Adverse Events (participants affected / at risk) | 32/130 | 21/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Zoster Vaccine (RZV) and Quadrivalent Adjuvanted Influenza Vaccine (N=130) | Recombinant Zoster Vaccine (RZV) and High-Dose Quadrivalent Influenza Vaccine (N=137)
Cardiovascular Accident (CVA), Unspecified Mechanism (Cardiac disorders) | 0 (0) | 1 (1)
Hepatocellular Carcinoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pulmonary embolism and acute deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Left partial cranial nerve III palsy (Nervous system disorders) | 0 (0) | 1 (1)
Revision of right shoulder rotator cuff surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalization for pacemaker due to arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (COPD) exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Zoster Vaccine (RZV) and Quadrivalent Adjuvanted Influenza Vaccine (N=130) | Recombinant Zoster Vaccine (RZV) and High-Dose Quadrivalent Influenza Vaccine (N=137)
COVID-19 Infection (Infections and infestations) | 15 (15) | 11 (11)
Upper Respiratory Infection (Infections and infestations) | 17 (17) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT05007041/Prot_003.pdf
  • Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT05007041/SAP_004.pdf
  • Informed Consent Form (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT05007041/ICF_000.pdf